CLINICAL TRIAL: NCT03935932
Title: Study of Humidified Air to Improve Mucociliary Clearance (MCC) in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frank C Sciurba (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor-Investigator, Frank C Sciurba, Professor of Medicine and Education, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19110243
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Results first posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: COPD
Keywords: COPD; Chronic bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic | interventions — Humidifiers

STUDY DESIGN:
Intervention Model Description: Open label, single treatment administration, crossover
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- baseline followed by intervention (Experimental): Subjects randomized to perform baseline measurement of clearance on study day 2 and measurement of clearance with nasal delivery of heated and humidified air on day 3
  Interventions: Device: nasal delivery of heated and humidified air
- intervention followed by baseline (Experimental): Subjects randomized to perform measurement of clearance with nasal delivery of heated and humidified air on day 2 and baseline measurement of clearance on study day 3
  Interventions: Device: nasal delivery of heated and humidified air

INTERVENTIONS:
Device: nasal delivery of heated and humidified air — Subjects will receive nasal delivery of heated and humidified air (plus oxygen if needed) at 30 liters/minute from the Fisher and Paykel myAirvo2 heater/humidifier using an Optiflow nasal cannula.
  Other Names: Fisher and Paykel myAirvo2 heater/humidifier; Optiflow nasal cannula.

SUMMARY:
This purpose of this study is to determine whether nasal delivery of heated and humidified air for a period of 4 hours will improve the clearance of mucus from the lungs of patients with chronic obstructive pulmonary disease (COPD). Mucus clearance will be measured using a nuclear medicine imaging procedure called a mucociliary clearance scan. Humidified air (with added oxygen if needed) will be delivered from the Fisher and Paykel myAirvo2 heater/humidifier through an Optiflow nasal cannula.

DETAILED DESCRIPTION:
Chronic bronchitis is a component of Chronic Obstructive Pulmonary Disease (COPD), along with emphysema. COPD is associated with smoking, exposure to environmental pollutants, or occupational exposures. In the airways mucus acts to trap inhaled toxins or pathogens. In a healthy lung mucus is cleared by mucociliary and cough clearance. Mucociliary clearance involves the synchronous motion of cilia underneath the mucus sheet that lines the airways. This drives the mucus sheet out of the airways (like a conveyer belt) continually clearing particulate and pathogens. In chronic bronchitis, mucus is overproduced due to toxic stimuli. Mucus clearance may also be defective due to airway obstruction and insufficient cough. This results in the accumulation of mucus that contributes to airway obstruction.

Therapies for improving mucus clearance may decrease the degree of airway obstruction experienced by COPD patients. Heated, high-flow, humidified air or oxygen may improve mucus clearance by hydrating the mucus in the airways and may also help to increase airway patency. A similar intervention was shown to improve mucus clearance in subjects with bronchiectasis.

The investigators have developed nuclear imaging-based methods for measuring mucus clearance from the lungs. These techniques have been applied to evaluate novel therapies for the treatment of cystic fibrosis lung disease. Here the investigators will apply these techniques to determine whether treatment with heated-humidified air will improve mucus clearance in subjects with COPD.

Study participation involves 3 visits.

Study day 1 includes:

1. A conversation with a physician and completion of informed consent
2. Pulmonary function testing (including albuterol administration)
3. The completion of a series of questionnaires

Study days 2 and 3 include:

1. A urine pregnancy test (if applicable)
2. Performance of a Co57 transmission scan
3. The inhalation of a radiopharmaceutical (Technetium-99m sulfur colloid) from a nebulizer
4. Lying flat in a nuclear medicine camera for 90 minutes while scans are collected.
5. Remaining at the test center for a follow up scan approximately 2.5 hours later. This scan will take 10 minutes.
6. Nasal delivery of heated humidified air (with supplemental oxygen if needed) at a rate of 30 liters per minute through a nasal cannula, on one study day. This will be started during the first 10 minutes of the 90 minute scanning period and continued for 4 hours. One the other study day there will be no treatment so that a baseline measurement of mucociliary clearance can be made. The order of the study days will be randomized.

Participants will be asked to refrain from using short-acting beta agonist (SABA) medications for 6 hours prior to study days 2 and 3, and long-acting beta agonists (LABA) or long-acting muscarinic antagonists (LAMA) for 24 hours prior to study days 2 and 3.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female 40 to 85 years old
2. Diagnosis of chronic bronchitis
3. Able to regularly produce sputum
4. Clinically stable
5. Current smoker or ex-smoker with a tobacco history of ≥10 pack-years (1 pack year = 20 cigarettes smoked per day for 1 year)
6. History of moderate to very severe COPD with a post-bronchodilator FEV1/FVC<0.70 and a post-bronchodilator FEV1>20% and ≤70% of predicted normal value at enrollment.
7. CAT score ≥ 10, with questions 1 and 2 responses ≥ 5

Exclusion Criteria:

1. Pregnant or nursing or unwilling to perform pregnancy testing
2. Unwilling or unable to refrain for SABA/LABA use ahead of the study
3. Unable to lie recumbent for 90 min,
4. Clinically important pulmonary disease other than COPD (e.g. active lung infection, clinically significant bronchiectasis, pulmonary fibrosis, cystic fibrosis, hypoventilation syndrome associated with obesity, lung cancer, alpha 1 anti-trypsin deficiency and primary ciliary dyskinesia) or another diagnosed pulmonary or systemic disease that is associated with elevated peripheral eosinophil counts (e.g. allergic bronchopulmonary aspergillosis/mycosis, Churg-Strauss syndrome, hyper-eosinophilic syndrome) and/ or radiological findings suggestive of a respiratory disease other than COPD that is contributing to the subject's respiratory symptoms.
5. Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric, or major physical impairment that is not stable in the opinion of the Investigator and/or could:

   * Affect the safety of the subject throughout the study
   * Influence the findings of the study or their interpretation
   * Impede the subject's ability to complete the entire duration of study
6. Treatment with systemic corticosteroids and/or antibiotics, and/or hospitalization for a COPD exacerbation within 2 weeks prior to enrollment, based on last dose of steroids or last date of hospitalization whatever occurred later
7. Acute upper or lower respiratory infection within 2 weeks prior to enrollment
8. Supplemental oxygen use at greater than 3 liters/min

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank C Sciurba, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Baseline Followed by Intervention: Subjects randomized to perform baseline measurement of clearance on study day 2 and measurement of clearance with nasal delivery of heated and humidified air on day 3. Study days are separated by 4-7 days
  nasal delivery of heated and humidified air: Subjects will receive nasal delivery of heated and humidified air (plus oxygen if needed) at 30 liters/minute from the Fisher and Paykel myAirvo2 heater/humidifier using an Optiflow nasal cannula for four hours
- Intervention Followed by Baseline: Subjects randomized to perform measurement of clearance with nasal delivery of heated and humidified air on day 2 and baseline measurement of clearance on study day 3. Study days are separated by 4-7 days.
  nasal delivery of heated and humidified air: Subjects will receive nasal delivery of heated and humidified air (plus oxygen if needed) at 30 liters/minute from the Fisher and Paykel myAirvo2 heater/humidifier using an Optiflow nasal cannula for 4 hours.
Period: Overall Study
Arm/Group | Baseline Followed by Intervention | Intervention Followed by Baseline
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baseline Followed by Intervention | Intervention Followed by Baseline | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [53 to 74] | 70 [62 to 75] | 70 [59 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Mucociliary Clearance Rate - 4 Hours
Description: Percentage of radioactivity cleared from the right lung
Time Frame: 0-4 hours
Measure: Median (Inter-Quartile Range); unit: percent clearance
Groups:
- AIRVO Day: Nasal delivery of heated and humidified air: Subjects will receive nasal delivery of heated and humidified air (plus oxygen if needed) at 30 liters/minute from the Fisher and Paykel myAirvo2 heater/humidifier using an Optiflow nasal cannula.
- Baseline Day: Baseline assessment of mucociliary clearance
Arm/Group | AIRVO Day | Baseline Day
Number analyzed (Participants) | 12 | 12
percent clearance | 47 [23 to 66] | 56 [40 to 68]
Statistical Analysis 1: Comparison: AIRVO Day vs Baseline Day; Test type: Other; p = 0.11, Wilcoxon signed-rank

2. Secondary Outcome: Mucociliary Clearance Rate - 90 Min
Description: Percentage of radioactivity cleared from the right lung
Time Frame: 0-90 minutes
Measure: Median (Inter-Quartile Range); unit: percent clearance
Groups:
- Baseline Day: Baseline measure of mucociliary clearance
Arm/Group | Airvo Day | Baseline Day
Number analyzed (Participants) | 12 | 12
percent clearance | 22 [14 to 31] | 34 [17 to 47]
Statistical Analysis 1: Comparison: Airvo Day vs Baseline Day; Test type: Other; p = 0.11, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Area Above Retention Curve - 90 Min
Description: Area above the curve of normalized retention of radioactivity vs time from the right lung
Time Frame: 0-90 minutes
Measure: Median (Inter-Quartile Range); unit: percent clearance x time (minutes)
Arm/Group | Airvo Day | Baseline Day
Number analyzed (Participants) | 12 | 12
percent clearance x time (minutes) | 6.2 [2.3 to 8.8] | 8.0 [1.4 to 11.9]
Statistical Analysis 1: Comparison: Airvo Day vs Baseline Day; Test type: Other; p = 0.35, Wilcoxon signed-rank

ADVERSE EVENTS:
Time Frame: study days only, up to14 days
Arm/Group | Airvo Day | Baseline Day
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Airvo Day (N=12) | Baseline Day (N=12)
flank pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
burning sensation in chest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT03935932/Prot_001.pdf
  • Statistical Analysis Plan (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/32/NCT03935932/SAP_003.pdf